CLINICAL TRIAL: NCT07188896
Title: A Randomized Phase 2 Trial of Fianlimab and Cemiplimab +/- Ipilimumab or Ipilimumab Plus Nivolumab in First-line Advanced Renal Cell Carcinoma (RCC)
Brief Title: A Randomized Trial of Fianlimab and Cemiplimab +/- Ipilimumab or Ipilimumab Plus Nivolumab in First-line Advanced Renal Cell Carcinoma (RCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brian Rini (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Brian Rini, Sponsor-investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU23-651
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Renal Cell Carcinoma (aRCC); Metastatic Renal Cell Carcinoma ( mRCC); Clear Cell Renal Cell Carcinoma (ccRCC)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab; Nivolumab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Cemiplimab, Fianlimab, and Ipilimumab (Experimental): Cemiplimab and fianlimab will be co-administered by IV. Ipilimumab will be administered by IV.
  Interventions: Drug: Fianlimab; Drug: Ipilimumab; Drug: Cemiplimab
- Arm B: Cemiplimab and Fianlimab (Experimental): Cemiplimab and fianlimab will be co-administered by IV.
  Interventions: Drug: Fianlimab; Drug: Cemiplimab
- Arm C: Nivolumab and Ipilimumab (Active Comparator): Nivolumab and ipilimumab will be by IV. Nivolumab will be administered by IV after the combination.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Fianlimab — Fianlimab will be co-administered by IV.
  Arms: Arm A: Cemiplimab, Fianlimab, and Ipilimumab; Arm B: Cemiplimab and Fianlimab
Drug: Ipilimumab — Ipilimumab will be administered by IV.
  Other Names: Yervoy
  Arms: Arm A: Cemiplimab, Fianlimab, and Ipilimumab; Arm C: Nivolumab and Ipilimumab
Drug: Nivolumab — Nivolumab will be administered by IV. Maintenance nivolumab will then be administered by IV.
  Other Names: Opdivo
  Arms: Arm C: Nivolumab and Ipilimumab
Drug: Cemiplimab — Cemiplimab will co-administered by IV.
  Arms: Arm A: Cemiplimab, Fianlimab, and Ipilimumab; Arm B: Cemiplimab and Fianlimab

SUMMARY:
This three-arm randomized phase 2 trial will enroll advanced clear cell RCC patients (all IMDC risk groups). Patients will be randomized 2:2:1 to either Arm A (fianlimab/ cemiplimab/ ipilimumab), Arm B (fianlimab/ cemiplimab), or Arm C (standard ipilimumab/ nivolumab), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Karnofsky Performance Status ≥ 70% within 14 days prior to registration.
4. Histological or cytological evidence of renal cell carcinoma having a clear cell component
5. Advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV [version 9]) renal cell carcinoma.
6. Treatment naïve for systemic therapy for renal cell carcinoma including no prior neo/adjuvant systemic therapy
7. Measurable disease according to RECIST 1.1 within 28 days prior to registration.
8. Patient must have either a formalin-fixed, paraffin-embedded (FFPE) tissue block or unstained tumor tissue sections, obtained from preferably a metastatic lesion, preferably within 3 months or no more than 12 months with an associated pathology report. If the metastatic lesion biopsy specimen does not contain at least 20 unstained slides, supplementation with primary kidney cancer tissue is acceptable.
9. Demonstrate adequate organ function as defined in the protocol. All screening labs to be obtained within 14 days prior to registration.
10. Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration.
11. Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from penile-vaginal intercourse or must use an effective method(s) of contraception. Males able to father a child who are sexually active with a female of childbearing potential must be willing to abstain from penile-vaginal intercourse or use an effective method(s) of contraception.
12. Known HIV-infected subjects on effective anti-retroviral therapy with undetectable viral load and CD4 count above 350 either spontaneously or on a stable antiviral regimen within 6 months of registration are eligible for this trial. Testing is not required at screening unless mandated by local policy
13. Subjects with known chronic hepatitis B virus (HBV) infection, must have an undetectable HBV viral load (serum hepatitis B virus DNA PCR that is below the limit of detection) and be on suppressive therapy, if indicated.
14. Subjects with a history of hepatitis C virus (HCV) infection must have been treated and cured (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy). For subjects with HCV infection who are currently on treatment, the HCV viral load must be undetectable to be eligible for this trial. Testing is not required at screening unless mandated by local policy.
15. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Prior systemic therapy against renal cell carcinoma in the neo/adjuvant or metastatic setting
2. Any condition requiring ongoing ≥ 10 mg prednisone equivalent/day
3. Participants with a history of myocarditis.
4. If clinically indicated based on clinical assessment and any ECG abnormalities, optional troponin T (TnT) or troponin I (TnI) may be done as described in the protocol.
5. Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are allowed: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
6. Central nervous system (CNS) metastases as described in the protocol.
7. Active infection requiring systemic therapy as described in the protocol.
8. Pregnant or breastfeeding as described in the protocol.
9. Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen, per treating physician discretion.
10. Subjects must not receive live attenuated vaccines within 4 weeks prior to Cycle 1 Day 1 or at any time during the study. Inactivated vaccines are allowed.
11. Known hypersensitivity to the active substances or to any of the excipients.
12. Currently participating in another study or participated in any study of an investigational agent or investigational device within 30 days of the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  ORR is defined as confirmed complete response (CR) + confirmed partial response (PR) and will be determined as per RECIST 1.1.

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) | 5 years
  PFS is defined as the time from Day 1 of treatment to the first documented disease progression per RECIST 1.1, clinically progressive disease per investigator, or death due to any cause, whichever occurs first.
12-month Progression Free Survival (PFS) | 12 months
  PFS is defined as the time from Day 1 of treatment to the first documented disease progression per RECIST 1.1, clinically progressive disease per investigator, or death due to any cause, whichever occurs first.
24-month Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from Day 1 of treatment to the first documented disease progression per RECIST 1.1, clinically progressive disease per investigator, or death due to any cause, whichever occurs first.
Duration of Response (DOR) | 5 years
  DOR is defined as the time from first documented evidence of CR or PR per RECIST 1.1 until disease progression based on RECIST 1.1 or death due to any cause, whichever occurs first.
Treatment Free Survival (TFS) | 5 years
  TFS will be assessed based on the area between two time to event KM curves from the time of study treatment initiation to study treatment discontinuation and from study initiation to initiation of subsequent systemic anti-cancer treatment or death. Time on or off treatment with Grade 3 or greater treatment related toxicities per CTCAE v5 will be determined as the area between study initiation and toxicity start and study initiation and Grade 3 toxicity ending.
Adverse Event Rates | 5 years
  The frequency of subjects experiencing treatment related adverse events and SAEs graded per NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center